CLINICAL TRIAL: NCT01646346
Title: A Pilot Study of Four-Dimensional Conformal Image Guided Accelerated Partial Breast Irradiation In The Treatment Of Stage 0 and l Breast Cancer
Brief Title: 4D Image-Guided Partial Breast Radiation in Stage 0 and l Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1110009173
Record Dates: First submitted 2012-03-11; First posted 2012-07-20 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Radiation for Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 4D Conformal Image-Guided Partial Breast RT (Experimental): This is a single arm trial designed to look at the results in women treated with partial breast irradiation twice daily for 5 days.
  Interventions: Radiation: 4D Conformal Image-Guided Partial Breast RT

INTERVENTIONS:
Radiation: 4D Conformal Image-Guided Partial Breast RT — External beam partial breast radiation to target a portion of the breast twice a day for 5 days.
  Other Names: 4D conformal image guided radiation therapy

SUMMARY:
The Purpose of this study is to evaluate the feasibility of using image guidance and four-dimensional computed tomography to reduce the volume of non target breast tissue that is treated with accelerated partial breast irradiation via the external beam technique.

DETAILED DESCRIPTION:
This is a pilot study enrolling about 30 patients to evaluate the feasibility of using 4D CT and daily image guidance in Accelerated Partial Breast Irradiation (APBI) to decrease set-up error and individualized planning target volumes to limit the non-target breast tissue dose. The two specific breasts constraints which shall be decreased are the V50 (percent volume of breast receiving 50% of the prescribed dose) and the V100 (percent volume of breast receiving 100% of the prescribed dose). The goal will be to decrease these to 45% and 23.5% respectively, which is down 33% from the NSABP B39 standard of 60% and 35%.

ELIGIBILITY:
Inclusion Criteria:

* The patient must consent to be in the study and must have a signed an approved consent form conforming with institutional guidelines.
* Patient must be > 50 years old.
* The patient should have a life expectancy of at least two years with a karnofsky performance status > 70.
* The patient must have stage 0 or I breast cancer.
* On histological examination, the tumor must be DCIS or invasive adenocarcinoma of the breast.
* Surgical treatment of the breast must have been lumpectomy. The margins of the resected specimen must be histologically free of tumor (>2mm, DCIS and invasive). Re-excision of surgical margins is permitted.
* Gross disease must be unifocal with pathologic (invasive and/or DCIS) tumor size 2 cm or less. (Patients with microscopic multifocality are eligible as long as total pathologic tumor size is 2 cm or less.)
* Patients with invasive breast cancer are required to have axillary staging which can include sentinel node biopsy alone (if negative), sentinel node biopsy followed by axillary dissection or sampling with a minimum total of 6 axillary nodes or axillary dissection alone (with a minimum of 6 axillary nodes). Axillary staging is NOT required for patients with DCIS.
* The patient must have simulation within 8 weeks/56 days of the final surgery for their breast cancer (lumpectomy, re-excision of margins, or axillary staging procedure).
* Patients with a history of non-ipsilateral breast malignancies are eligible if they have been disease-free for 2 or more years prior to enrollment. Patients with the following cancers are eligible even if diagnosed and treated within the past 2 years: carcinoma in situ of the cervix, colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Chemotherapy is permitted if planned for ≥ 2 weeks after radiation.
* Urine pregnancy test must be performed and be negative on all women younger than 60 who have not had a tubal ligation, oophorectomy, or hysterectomy.
* Separate incisions for the lumpectomy and sentinel node biopsy should be present. Use of only one incision will typically result in a contiguous cavity with the tumor bed and the sentinel node sampling, and inability of the radiation oncologist to delineate the tumor bed from the sentinel node bed.
* The patient must have a cavity which is able to be targeted with external beam APBI, either through surgical clip placement, or CVS 3 or higher. The cavity to whole breast ratio must be 30% or less.

Exclusion Criteria:

* Men are not eligible for this study as men are not breast conservation candidates.
* T0, T2 (> 2.0 cm), T3, node positive, stage III or IV breast cancer.
* Any positive axillary nodes.
* Palpable or radiographically suspicious ipsilateral or contralateral axillary, supraclavicular, infraclavicular or internal mammary nodes, unless biopsy proven to be negative for tumor.
* Suspicious microcalcifications, densities or palpable abnormalities in either breast unless biopsy proven to be benign.
* Non-epithelial breast malignancies such as sarcoma or lymphoma.
* Proven multicentric carcinoma in more than one quadrant or separated by more than 2 centimeters.
* Paget's disease of the nipple.
* History of invasive breast cancer or DCIS in the same breast.
* Surgical margins that cannot be microscopically assessed or are less then 2 mm.
* Collagen vascular disease, specifically dermatomyositis with a CPK level above normal or with an active skin rash, systemic lupus erythematosis or scleroderma.
* Pregnancy or lactation at the time of proposed radiation. Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the treating physician, would preclude the patient from meeting the study requirements.
* Patients with coexisting medical conditions in whom life expectancy is < 2 years.
* Patients with skin involvement, regardless of tumor size.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-01-10 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Evans, MD, Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Hospital Care Center, Yale New Haven Hospital, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 54 people were recruited to take part, however only 46 of those were treated and included in the study.
Period: Overall Study
Arm/Group | 4D Conformal Image-Guided Partial Breast RT
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 4D Conformal Image-Guided Partial Breast RT
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 64.0 [50 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Patients With Reduction in Incidental Radiation
Description: Patients were assessed to determine if there was a reduction in breast radiation V50 less than 45% and V100 less than 23.5%.
Time Frame: 5 day
Measure: Count of Participants; unit: Participants
Arm/Group | 4D Conformal Image-Guided Partial Breast RT
Number analyzed (Participants) | 46
Participants | 46

2. Secondary Outcome: Cosmesis by Patient Report
Description: This outcome is measured by the Breast Cancer Treatment outcome Scale (BCTOS). Eleven items (e.g., breast size, breast pain, breast shape) are rated by patients on a 4-point scale (0=no difference to 3=large difference), with a score range of 0-33 (higher scores signifying worse outcome). Scores on each item are summed to obtain a total score.
Time Frame: Within no more than 8 weeks of surgery, but prior to the start of radiation
Measure: Median (Full Range); unit: units on a scale
Arm/Group | 4D Conformal Image-Guided Partial Breast RT
Number analyzed (Participants) | 46
units on a scale | 4 [0 to 16]

3. Secondary Outcome: Cosmesis by Patient Report
Description: as for outcome 2
Time Frame: 1 year post treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | 4D Conformal Image-Guided Partial Breast RT
Number analyzed (Participants) | 43
units on a scale | 8.5 [1 to 20]

4. Secondary Outcome: Cosmesis by Patient Report
Description: as for outcome 2
Time Frame: 3 year post treatment
Measure: Median (Full Range); unit: units on a scale
Arm/Group | 4D Conformal Image-Guided Partial Breast RT
Number analyzed (Participants) | 39
units on a scale | 7.0 [0 to 29]

5. Secondary Outcome: Cosmesis by Medical Doctor Report
Description: Medical doctor will be provided with cosmesis scale and grade cosmesis of breast. Cosmesis was based on the Harvard Cosmesis Scale rated as :1. excellent: the treated breast looked essentially the same as the opposite breast; 2. good: minimal but identifiable effects of radiation on the treated breast; 3. fair: significant effects of radiation on the breast were noted; 4. severe normal tissue sequelae.
Time Frame: Within no more than 8 weeks of surgery, but prior to the start of radiation
Measure: Count of Participants; unit: Participants
Arm/Group | 4D Conformal Image-Guided Partial Breast RT
Number analyzed (Participants) | 46
Participants
  excellent | 41
  good | 4
  fair | 1
  poor | 0

6. Secondary Outcome: Cosmesis by Medical Doctor Report
Description: as for outcome 5
Time Frame: 1 yr post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 4D Conformal Image-Guided Partial Breast RT
Number analyzed (Participants) | 43
Participants
  excellent | 20
  good | 20
  fair | 3
  poor | 0

7. Secondary Outcome: Cosmesis by Medical Doctor Report
Description: as for outcome 5
Time Frame: 3 yr post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | 4D Conformal Image-Guided Partial Breast RT
Number analyzed (Participants) | 39
Participants
  excellent | 16
  good | 17
  fair | 5
  poor | 1

ADVERSE EVENTS:
Time Frame: Through treatment completion, and up to 3 years follow up.
Arm/Group | 4D Conformal Image-Guided Partial Breast RT
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 45/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4D Conformal Image-Guided Partial Breast RT (N=46)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 14 (15)
General disorders and administration site conditions (General disorders) | 1 (1)
Localized edema (General disorders) | 14 (15)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 2 (3)
Dermatitis radiation (Injury, poisoning and procedural complications) | 25 (31)
Seroma (Injury, poisoning and procedural complications) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Superficial soft tissue fibrosis (Injury, poisoning and procedural complications) | 41 (57)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 13 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fat atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 5 (7)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 38 (51)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 4 (4)
Telangiectasia (Skin and subcutaneous tissue disorders) | 5 (6)
Thromboembolic event (Vascular disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT01646346/Prot_SAP_000.pdf